CLINICAL TRIAL: NCT05662787
Title: BOLT Lithotripsy RESTORE ATK Trial for PAD (RESTORE ATK)
Brief Title: BOLT Lithotripsy RESTORE ATK Trial
Acronym: RESTORE ATK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bolt Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-001701
Record Dates: First submitted 2022-11-30; First posted 2022-12-23 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, non- randomized, multi-center study for treatment of stenotic lesions with the Bolt Intravascular Lithotripsy system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intravascular lithotripsy (Experimental)
  Interventions: Device: Intravascular Lithotripsy

INTERVENTIONS:
Device: Intravascular Lithotripsy — Enhancing percutaneous transluminal angioplasty by utilizing delivery of IVL to disrupt calcium in above the knee lesions prior to full balloon dilatation at low pressures

SUMMARY:
The RESTORE (ATK) above the knee study is a prospective, non- randomized, multi-center study for treatment of stenotic lesions with the Bolt Intravascular Lithotripsy System.

DETAILED DESCRIPTION:
The RESTORE (ATK) above the knee study is a prospective, non- randomized, multi-center study for treatment of stenotic lesions with the Bolt Intravascular Lithotripsy System that was designed to enhance percutaneous transluminal angioplasty by utilizing delivery of intravascular lithotripsy (IVL) to disrupt calcium prior to full balloon dilatation at low pressures.

ELIGIBILITY:
Inclusion Criteria:

* Age of subject is ≥18.
* Rutherford Clinical Category 2, 3, or 4.
* Target lesion that is located in a native de novo superficial femoral artery (SFA) or popliteal artery (popliteal artery extends to and ends proximal to the ostium of the anterior tibial artery)
* Calcification is at least moderate. (presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending ≥ 50% the length of the lesion or absolute length ≥20mm.

Exclusion Criteria:

* Planned major amputation of the target leg (above the ankle)
* The use of chronic total occlusion (CTO) re-entry devices
* CTOs greater than 80 mm in length
* Lesions within 10 mm of ostium of the SFA
* Significant stenosis (>50% stenosis) or occlusion of inflow tract before target treatment zone (e.g., iliac or common femoral) not successfully treated with percutaneous angioplasty (PTA) or stent and without complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | Immediately after the intervention/procedure/surgery
  Post-treatment residual diameter stenosis of < 50% of the target lesion (with or without adjunctive PTA therapy and/or stenting)
Primary Safety Endpoint | Within 30 days following procedure
  Composite of New-onset Major Adverse Events (MAEs)

SECONDARY OUTCOMES:
Freedom from Major Adverse Events (MAEs) within 6 months. | Within 6 months following procedure
  Freedom from MAE within 6 months
Residual diameter stenosis of <50% of the target lesion (without adjunctive PTA or stent therapy) | Immediately after the intervention/procedure/surgery
  Residual diameter stenosis of <50% of the target lesion (without adjunctive PTA or stent therapy)
Residual diameter stenosis of <30% of the target lesion (without adjunctive PTA or stent therapy) | Immediately after the intervention/procedure/surgery
  Residual diameter stenosis of <30% of the target lesion (without adjunctive PTA or stent
Target lesion patency - freedom from > 50% restenosis (assessed by DUS) | 30 days following procedure
  Target lesion patency - freedom from > 50% restenosis (assessed by DUS)
Target lesion patency - freedom from > 50% restenosis (assessed by DUS) | 6 months following procedure
  Target lesion patency - freedom from > 50% restenosis (assessed by DUS)
Freedom from Target Lesion Revascularization (TLR) at 6 months | 6 months following procedure
  Freedom from Target Lesion Revascularization (TLR) at 6 months
Ankle-Brachial Index (ABI) of the target limb at all planned follow-up time points | at discharge after index procedure, 30 days following procedure, 6 months following procedure
  Ankle-Brachial Index (ABI) of the target limb at all planned follow-up time points

CONTACTS AND LOCATIONS:
Locations (10):
- Austria (3):
  - Medical University of Graz, Graz
  - Universitätsklinik für Innere Medizin II, Vienna
  - Mein Hanusch Krankenhaus, Vienna
- University Hospital of Split, Split, Croatia
- Germany (6):
  - Klinikum Hochsauerland GmbH, Arnsberg
  - Universitätsklinikum Freiburg Universitäts-Herzzentrum, Bad Krozingen
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Universitätsklinikum Münster (UKM), Münster
  - St. Franziskus-Hospital GmbH, Münster
  - GRN Klinik Weinheim, Weinheim